CLINICAL TRIAL: NCT04678466
Title: An Expanded Access Program Providing Flotetuzumab in the Treatment of Acute Myeloid Leukemia Patients in Single, Individually-approved Patients
Brief Title: Flotetuzumab Expanded Access Program
Status: No longer available | Type: Expanded Access
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Other Study IDs: MGD006-EA
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Acute Myeloid Leukemia; AML; AML, Adult Recurrent
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: flotetuzumab — CD123 x CD3 bispecific DART® antibody
  Other Names: MGD006

SUMMARY:
The purpose of the Expanded Access program is to provide flotetuzumab to patients with acute myeloid leukemia (AML) for whom potential benefit justifies potential treatment risks.

DETAILED DESCRIPTION:
MacroGenics will consider, on a case-by-case basis, requests by treating physicians to file a single patient investigational new drug application for expanded access to flotetuzumab and for MacroGenics to supply flotetuzumab for single patient use.

ELIGIBILITY:
Inclusion Criteria:

* Weight of at least 17 kilograms
* CD123-positive hematologic malignancy
* Adequate organ reserve
* Provider and site are trained on study protocol using flotetuzumab

Exclusion Criteria:

* AML that meets inclusion criteria for study CP-MGD006-01 (NCT02152956)
* Primary induction failure
* Early relapse (less than 6 months after first complete remission )
* Three prior lines of therapy, including maximum of 1 prior salvage attempts

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Ward, MD, Study Director — MacroGenics